CLINICAL TRIAL: NCT05363813
Title: Post-market Clinical Follow-up Study of REusable Clip Applier and Cartridge Devices for LAParoscopic Surgery
Brief Title: Post-market Clinical Follow-up Study of Reusable Clip Applier Cartridge Devices for LAParoscopic Surgery
Acronym: RELAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microline Surgical, Inc. (Industry)
Collaborators: AKRN Scientific Consulting, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD01-227
Record Dates: First submitted 2022-04-28; First posted 2022-05-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Minimally Invasive Surgical Procedures; Laparoscopy; Leakage of Cardiac Device
Keywords: Laparoscopy; PMCF; Laparoscopic surgery; Vessel ligation; Duct ligation; Vessel leakage; Duct leakage

STUDY DESIGN:
Intervention Model Description: Patient selection based on need for laparoscopic surgical treatment involving vessel or duct ligation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Laparoscopic Surgical Patients (Experimental): 1. Adult subjects, male or female, ≥18 years old
  2. Subjects who have been scheduled for a laparoscopic surgery using the clip
  3. Subjects who had provided written informed consent form
  4. Ability and willingness to comply with all study requirements to be evaluated for each study visit
  Interventions: Device: M/L-10 Multi-Fire Clip Applier and M/L-10 Clip Cartridge (Multi-Fire Clip System)

INTERVENTIONS:
Device: M/L-10 Multi-Fire Clip Applier and M/L-10 Clip Cartridge (Multi-Fire Clip System) — Permanent ligation of vessels and ducts as part of minimally invasive laparoscopic surgery.

SUMMARY:
This is a Post-Market Clinical Follow-up (PMCF) investigation to determine the long-term effectiveness and safety of the Multi-Fire Clip System in laparoscopic surgery. This system consists of two medical devices, the M/L-10 Clip Applier and the M/L-10 Clip. The Multi-Fire Clip System is indicated for occluding and ligating vessels, ducts, tracts and other tubular structures during laparoscopic and general surgical procedures. This medical device has been marketed in Europe since 2006 and in the United States since 2002, among other places.

Laparoscopic surgeries have become the standard of excellence for many surgical procedures as they allow the intervention to be performed in a minimally invasive way, which means significant improvements in factors such as postoperative pain or length of hospital stay compared to open surgeries. Laparoscopic procedures require the use of different hemostatic techniques to minimize blood loss or leakage of other fluids through their respective ducts. Currently, clip and staple placement are the most commonly used procedures for ligation and/or occlusion of blood vessels and other tubular structures.

In this context, the Multi-Fire Clip System is presented as an alternative device that can produce significant cost savings due to the reusable design of the M/L-10 Clip Applier. It also provides precise control of bleeding during surgery, which could lead to less potential injury to surrounding structures.

The present clinical trial is a PMCF study to evaluate the long-term safety and efficacy of the Multi-Fire Clip System in patients scheduled to undergo laparoscopic surgery in which clip placement is anticipated. During the surgery procedure, the necessary clips will be placed using the aforementioned multi-shot clip system. Participants will be followed up for 6 months after the operation. Through an on-site visit and a telephone call visit, data on possible adverse events related to the device or procedure will be collected in order to assess the long-term safety and efficacy of these devices.

DETAILED DESCRIPTION:
The RELAP PMCF will be conducted as a prospective, single-arm, open-label and multi-center clinical investigation and will include up to 230 subjects derived for laparoscopic surgery. The clinical investigation will be conducted in up to 12 sites located in European countries. Additional sites or other countries may be approached for participation in the clinical investigation if needed.

The primary objective of the RELAP Post-Market Clinical Follow-Up Study is to determine the long-term effectiveness of the Multi-Fire Clip System through 6-months follow-up. The secondary objective of the RELAP Post-Market Clinical Follow-Up Study is focused on the long-term evaluation of Multi-Fire Clip System safety and effectiveness through the collection of Serious Adverse Events (SAEs) and Major Adverse Events (MAEs) related to both the medical device and the procedure.

The primary safety and efficacy endpoint is the efficacy of long-term vessel/duct ligation defined as absence of Adverse Events (AEs) related to vessel and/or duct leakage due to incomplete ligation of the vessel/duct after appropriate placement of clip at 6 months in patients indicated for laparoscopic surgical procedure.

There are several secondary endpoints planned for his clinical investigation. Firstly, all serious adverse events (SAEs) will be evaluated at 6 months. Additionally, a long-term evaluation of major adverse events (MAEs) related to both the medical device and the procedure. A Risk Ratio (RR) will be defined for the analysis of this secondary endpoint. The time frame for the long-term evaluation will be 30-days follow-up and 6-months follow-up. Moreover, the Acute Procedural Success (APS), defined as the absence of (S)AEs within 24h after the surgery, will be assessed. The Acute Device Success, defined as the absence of (S)AEs related to the devices within the 24h after the surgery will also be evaluated. Finally, the Length of Stay (LoS) in the hospital will be evaluated.

The Clinical Investigation visits will occur at Baseline, Procedure and 30-days follow-up, with a final phone call at 6 months will take place. This clinical investigation will enroll male and female adult subjects who have been scheduled for a laparoscopic surgery using a clip. Subjects must meet all eligibility criteria and provide written informed consent prior to conducting any investigation-specific procedures not considered standard of care. The target population are subjects that require a laparoscopic surgery and a clip can be used to occlude a vessel/duct. Approximately 230 subjects will be enrolled in the clinical investigation in order to assess the primary endpoint. The expected duration of enrollment is up to 12 months. The expected duration of each subject's participation is 6 months, including the scheduled visits and data collection for this clinical investigation that will occur during the "early follow-up visit" at 30 days after the procedure and 6 months. The subject follow-up will be considered completed at the conclusion of their 6-month follow-up visit. Therefore, the total duration of the clinical investigation is expected to be 18 months.

Regarding the statistical analysis, the primary safety and effectiveness endpoint results will be compared with the data reported in the literature for similar medical devices. The analysis population will be the per-protocol (PP) population, and the results will be presented as the incidence (in percentage) of AEs related to leakage, with a 95% confidence. Further analyses using the PP population will be performed in order to verify the statistical robustness of the results. Secondary endpoints of this clinical investigation will refer to the assessment of the safety of laparoscopic surgical procedures through the collections of all SAEs reported at 6 months. In all cases, the PP population will be the analysis population, and results will be presented as a percentage, defining a Risk Ratio (RR), with 95% confidence. Other secondary endpoints of this clinical investigation include the acute device success and acute procedural success, which will be assessed during procedure. Besides, the length of hospital stay will also be analyzed, and data will be presented as total number of days.

The sample size calculation is based on the purpose to demonstrate non-inferiority of Multi-Fire Clip System compared to other metallic clips in terms of AEs related to fluid leakage. This assessment will allow to define a success rate of the long-term effectiveness and safety of M/L-10 Multi-Fire Clip System.

Primary data collection based on source-documented hospital and/or clinic chart reviews will be performed clearly and accurately by site personnel trained on the Clinical Investigation Plan (CIP) and Case Report Form (CRF) completion. The investigator will ensure accuracy, completeness, legibility and timeliness of the data reported to the Sponsor on the CRFs and in all required reports. Data on CRFs will be collected for all subjects that are enrolled into the clinical investigation. A Data Management Plan (DMP) will describe procedures used for data entry and collection. Data review and data cleaning, and issuing, resolving data discrepancies and methods for data base lock. The DMP will include procedures for the verification, validation and securing of electronic clinical system. The investigator/site will permit direct access to source data/documents for the purpose of performing clinical investigation-related monitoring, audits, EC review and regulatory inspections. Regulations and GCP require the Investigator to maintain information in the subject's original medical records that corroborates data collected on the CRFs. In order to comply with these regulatory requirements/GCP, medical history data, adverse events reported and their resolution as well as any other data required to substantiate data entered into the CRF, will be recorded. Data on CRFs will be collected for all subjects that are enrolled into the clinical investigation.

Sponsor and/or designee will monitor the clinical investigation over its duration according to the CIP-specific monitoring plan which will include the planned extent of source data verification. This monitoring plan will be a separate document that can be updated during the course of the study. As for the safety monitoring, Measures taken to avoid bias related to safety includes 100% of source data verification related to AEs documented in the Monitoring Plan. A Sponsor representative or designee may request access to all clinical investigation records, including source documentation, for inspection during a Quality Assurance audit.

This clinical investigation, sponsored by Microline Surgical Inc. (Beverly, USA), will be conducted in accordance with this CIP. All investigators involved in the conduct of the clinical investigation will be qualified by education, training, or experience to perform their tasks and this training will be documented appropriately.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, male or female, ≥18 years old
2. Subjects who have been scheduled for a laparoscopic surgery using the clip
3. Subjects who had provided written informed consent form
4. Ability and willingness to comply with all study requirements to be evaluated for each study visit

Exclusion Criteria:

1. Subjects referred for laparoscopic surgeries to reinforce a staple line or produce partial vessel occlusion
2. Significant surgical contraindications evaluated using the GOALS score
3. Subjects unsuitable for laparoscopic surgery according to PI discretion
4. Subjects who have coagulopathy or uninterruptible anticoagulation therapy
5. Subjects currently under steroid treatment
6. Subject has known allergy to device components (i.e., titanium, stainless steel)
7. Subjects who are participating in another trial which may affect the outcomes data on this study
8. Inability to adhere to study-related procedures
9. Subjects that require emergency surgeries associated with trauma and/or sepsis with a SOFA score ≥ 2 and/or septic shock should be excluded
10. Pregnant or lactating women at the time of the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Long-Term Ligation Performance | 6 months after laparoscopic surgical procedures
  Efficacy of long-term vessel/duct ligation defined as absence of Adverse Events (AEs) related to vessel and/or duct leakage due to incomplete ligation of the vessel/duct after appropriate placement of clip at 6 months of laparoscopic surgical procedures.

SECONDARY OUTCOMES:
All Serious Adverse Events (SAEs) | 30 days follow-up, and 6 months follow-up after laparoscopic surgical procedures
  SAEs are Adverse Events (AEs) that meet any of the criteria below:
  1. Led to a death,
  2. Led to a serious deterioration in health of the subject, that either resulted in
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient hospitalization or prolongation of existing hospitalization, or
     4. medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
     5. chronic disease
Long-term evaluation of Major Adverse Events (MAEs) related to the medical device | 30-days follow-up, and 6-months follow-up
  MAEs are adverse events that can occur due to the operative procedure include, but are not limited to:
  * Major bleeding requiring reoperation
  * Septic shock from intraabdominal infection
  * Bowel injury requiring repair
  * Vascular injuries requiring repair
  * Genitourinary injuries requiring repair
  * Biliary injuries requiring repair
  * Retained foreign body, which is a patient safety incident in which a surgical object is accidentally left in a body cavity or operation wound following a procedure.
  MAES can also occur due to Anesthesia include, but are not limited to:
  * Cerebrovascular Accident (Stroke)
  * Myocardial Infarction
  * Pulmonary Embolism (PE)
  * Blood clots
  A Risk Ratio (RR) will be defined for the analysis of this secondary endpoint.
Long-term evaluation of Major Adverse Events (MAES) related to the procedure | 30-days follow-up, and 6-months follow-up
  MAEs are adverse events that can occur due to the operative procedure include, but are not limited to:
  * Major bleeding requiring reoperation
  * Septic shock from intraabdominal infection
  * Bowel injury requiring repair
  * Vascular injuries requiring repair
  * Genitourinary injuries requiring repair
  * Biliary injuries requiring repair
  * Retained foreign body, which is a patient safety incident in which a surgical object is accidentally left in a body cavity or operation wound following a procedure.
  MAES can also occur due to Anesthesia include, but are not limited to:
  * Cerebrovascular Accident (Stroke)
  * Myocardial Infarction
  * Pulmonary Embolism (PE)
  * Blood clots
  A Risk Ratio (RR) will be defined for the analysis of this secondary endpoint.
Acute Procedural Success (APS) | One day (during procedure)
  APS is defined as the absence of (S)AEs within 24h after the surgery.
Acute Device Success (ADS) | One day (during procedure)
  ADS is defined as the absence of (S)AEs related to the clip applier within 24h after the surgery.
Length of Stay (LoS) in hospital | Up to 30 days
  Patient's length of Stay (LoS) in hospital after laparoscopic surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Morales Conde, MD, Principal Investigator — Hospital QuirónSalud Sagrado Corazón, Sevilla, Spain
Locations (7):
- Centro Hospitalar Universitário Lisboa Norte, Lisbon, Portugal
- Spain (6):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruña del Área Sanitaria de A Coruña y Cee, A Coruña
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No